CLINICAL TRIAL: NCT02052817
Title: Randomized, Prospective Evaluation of the Toad Brace in Plantar Ulcer Off-loading and Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toad Medical Corporation (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Toad_Brace_07-13-11
Record Dates: First submitted 2014-01-20; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Foot; Pedal Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Debridement and standard of care in off-loading on control patients
  Interventions: Other: Optimal Medical Therapy - Debridement
- Toad Brace (Experimental): Debridement and fitting of Toad Brace
  Interventions: Device: Optimal Medical Therapy Debridement + Toad Brace

INTERVENTIONS:
Device: Optimal Medical Therapy Debridement + Toad Brace
  Arms: Toad Brace
Other: Optimal Medical Therapy - Debridement
  Arms: Control

SUMMARY:
The TOAD Medical Corporation Brace is a novel device that completely off-loads the foot and has been shown to heal ulcers at a rapid rate in preliminary experience in patients with plantar ulcers. This trial will attempt to show the efficacy of the Toad Brace and is based on the hypothesis that the Toad brace completely offloads the foot and hastens healing rates of diabetic ulcers. The trial will randomize 74 patients with diabetic pedal ulcers to the Toad Brace or conventional therapy. . Quantitative assessment of ulcer rate healing rates will be determined clinically and by blinded, computer-assisted planimetry of digital images over a 12 week period. The pressure on the plantar surface will be measured via a pressure sensor in a subset of patients. The trials will attempt to show markedly reduced pressure on the plantar surface and significantly higher ulcer healing rates with using the Toad Brace.

ELIGIBILITY:
Inclusion Criteria:

* Men or women >18 years old
* One or more foot ulcers without clinical evidence of osteomyelitis
* Diagnosis of Diabetes Mellitus*
* University of Texas Grade 1A, 1C, 2A, or 2C ulcer15
* ABI >0.7 and Toe pressure >30mmHg

Exclusion Criteria:

* Limited life-expectancy
* Wounds on calf or shin that would be in contact with the TAG Brace
* Gangrene, active infection
* Osteomyelitis of the foot with the ulcer
* Chronically bedridden/Non ambulatory
* Unable to keep research appointments
* Wide spread malignancy or systemically immunocompromising disease
* Ipsilateral revascularization procedure within the last 30 days.
* Unreliable, unwilling or unable to comprehend informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline measured wound area | Every 3 weeks for a period of 12 weeks
  We are taking repeated measures of wound area healing for pedal ulcers over a period of 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- UH Hospitals of Cleveland d/b/a University Hospitals Case Medical, Cleveland, Ohio, United States